CLINICAL TRIAL: NCT00205309
Title: Respiratory Tract IgA Levels in Critically Ill Intubated Patients
Brief Title: Airway IgA: Respiratory Tract IgA Levels in Critically Ill Intubated Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2002-562
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Intubation; Critically Ill
Keywords: intubated patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine the impact of acute illness on sequential airway IgA levels in intensive care patients who will require prolonged intubation. Infections are the most common cause of late deaths in non-head injured trauma patients and a frequent cause of morbidity and mortality in hospitalized patients, especially intubated Intensive Care Unit (ICU) patients. Nosocomial pneumonia is the most common of these infections, and its incidence in defined populations of critically injured patients is responsive to route and type of nutrition. This study will focus on the mechanisms of specific immune mucosal defenses in intestinal and extraintestinal sites and link enteral feeding (or lack of it) with maintenance (or deterioration) of respiratory mucosal defenses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be intubated, intensive care patients.

Exclusion Criteria:

* No severe pulmonary contusions or evidence of airway bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2003-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kudsk, MD, Principal Investigator — University of Wisconsin Medical School
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States